CLINICAL TRIAL: NCT05027854
Title: Brain Network Mechanisms Causally Underlying Human Decisions Revealed by Brain Stimulation and Functional MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Christian Ruff (Other)
Responsible Party: Sponsor-Investigator, Christian Ruff, Prof. Dr., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-01490
Record Dates: First submitted 2021-08-16; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Behavior and Behavior Mechanisms
MeSH Terms: conditions — Behavior | interventions — TES

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation (Experimental): TMS or tES, depending on experiment
  Interventions: Other: TMS or tES
- Sham (Sham Comparator): Corresponding sham TMS or tES
  Interventions: Other: sham TMS or tES

INTERVENTIONS:
Other: TMS or tES — Transcranial magnetic or electric stimulation
  Arms: Stimulation
Other: sham TMS or tES — Sham transcranial magnetic or electric stimulation
  Arms: Sham

SUMMARY:
We will examine how stimulation of specific brain areas with transcranial magnetic stimulation (TMS) or transcranial electric stimulation (tES) changes specific aspects of behavior and brain activity, in order to test hypotheses about brain behavior relationships (basic research).

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 80 years of age (whereby for most studies the majority of recruited participants will be between 18 and 40 years of age)
* right-handedness and/or one specific gender (male or female) can be inclusion criteria to reduce variation in the data.

Exclusion Criteria:

* inability to understand the instructions and insufficient knowledge of the project language
* Internal electronic and/or metallic objects in the head, neck, or shoulders (e.g. artificial cochleae, deep brain stimulators, medical pumps, shrapnel, metallic splinters due to accidents during metal welding)
* One or more epileptic fits in the participant or a first-degree relative
* Vascular, traumatic, tumoral, infectious, or metabolic brain damage
* Use of medication that significantly alters cortical excitability
* Acute sleep deprivation or withdrawal from alcohol
* pregnancy
* to reduce bias, students of psychology or economics can be excluded if there is a possibility that they are familiar with the relevant paradigm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Speed of Behaviour | 0-60 minutes after stimulation
  Reaction time in miliseconds
Accuracy of Behaviour | 0-60 minutes after stimulation
  Accuracy in percent correct
Cognitive Function driving Behaviour | 0-60 minutes after stimulation
  Parameter of Model describing cognitive function governing behaviour
Brain activity | 0-60 minutes after stimulation
  BOLD contrast in fMRI data

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ruff, PhD, Principal Investigator — University of Zurich

IPD SHARING:
Plan to Share IPD: Undecided